CLINICAL TRIAL: NCT01804634
Title: A Phase II Trial of Reduced Intensity Conditioning and Partially HLA-mismatched (HLA-haploidentical) Related Donor Bone Marrow Transplantation for High-risk Solid Tumors
Brief Title: Reduced Intensity Haploidentical BMT for High Risk Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J12106; NA_00076243 (Other: JHM IRB); 5P01CA225618-06 (NIH)
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Refractory and/or Relapsed Metastatic Solid Tumors
Keywords: Solid Tumors; Neuroblastoma; Osteosarcoma; Ewing Sarcoma; Rhabdomyosarcoma; Hepatoblastoma; Desmoplastic Round Cell Tumor
MeSH Terms: conditions — Neuroblastoma; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Hepatoblastoma | interventions — Cyclophosphamide; fludarabine; Influenza Vaccines; Whole-Body Irradiation; Melphalan; Honey; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced intensity conditioning (Experimental): Fludarabine IV infusion over 30 minutes on D-7 to D-3. The dose will be 30 mg/m2/dose (adjusted for renal function). Melphalan: IV infusion over 30-60 minutes, depending on volume, on D-2. The dose will be 100mg/m2.Total body irradiation: 200 cGy AP/PA with 4MV or 6MV photons at 8 12 cGy/min at the point of prescription (average separation of measurements at mediastinum, abdomen, and hips) will be administered in a single fraction on day -1. Bone Marrow will be harvested and infused on day 0. Post-transplantation Cyclophosphamide 50mg/kg will be given on D+3 post-transplant (within 60-72 hr of marrow infusion) and on D+4 post-transplant. Tacrolimus begins on Day 5, at least 24 hours after completion of posttransplantation Cy at 0.015mg/kg IBW/dose IV over 3 hours every 12 hours. Mycophenolic acid mofetil (MMF) F will be given at a dose of 15 mg/kg PO TID (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1 g PO TID).
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: low dose total body irradiation; Drug: Melphalan; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide — preparative regimen
  Other Names: cytoxan
Drug: Fludarabine
  Other Names: Flu
Radiation: low dose total body irradiation
  Other Names: TBI
Drug: Melphalan
  Other Names: Mel
Drug: Tacrolimus
  Other Names: tacro

SUMMARY:
The purpose of this study is to see if giving reduced intensity chemotherapy, haploidentical bone marrow, post-transplant cyclophosphamide and shortened duration tacrolimus is safe and feasible for patients with very high-risk solid tumors.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) may be associated with a clinically significant "graft-versus-tumor" (GVT) effect, even against disease that is unresponsive to chemotherapy and radiation therapy. Graft-vs.-tumor (GVT) effects have been described after allogeneic HCT for neuroblastoma, Ewing sarcoma, osteosarcoma, rhabdomyosarcoma, melanoma and hepatoblastoma.

The investigators' goal is to maximize a T cell and NK cell mediated graft versus tumor effect in poor prognosis solid tumor patients using haploidentical donors, T cell replete bone marrow, and a unique post-transplant immunosuppression regimen containing post transplantation Cy and shortened duration tacrolimus. This therapy will be widely applicable because almost all patients have a half-matched donor available (parent or sibling). The investigators hope to demonstrate the safety and feasibility of this therapy in anticipation of combining this platform with additional post-transplantation relapse/progression prevention therapy such as an immune checkpoint inhibitor.

TREATMENT PLAN Indwelling central venous catheter Placement of a double lumen central venous catheter will be required for administration of IV medications and transfusion of blood products.

Pre-treatment Evaluation All patients will require documentation of a detailed history and physical examination and standard evaluation of cardiac, pulmonary, liver and renal function. All patients will undergo disease evaluation as specified in Table 1, utilizing whichever modalities following the guidelines in 6.1.3 (i). Pre-BMT blood will be drawn per section section 5.12 for correlative labs.

Preparative regimen Fludarabine: administered as an IV infusion over 30 minutes on D-7 to D-3. The dose will be 30 mg/m2/dose (adjusted for renal function).

Melphalan: Recommended to be administered as an IV infusion over 30-60 minutes, depending on volume, on D-2. The dose will be 100mg/m2. Other institutional infusion standards are acceptable and will not be a protocol deviation.

Total body irradiation: 200 cGy AP/PA with 4MV or 6MV photons at 8 12 cGy/min at the point of prescription (average separation of measurements at mediastinum, abdomen, and hips) will be administered in a single fraction on day -1.

Day of rest: A day of rest, i.e. after preparative regimen completion and prior to bone marrow infusion, is not routinely scheduled. Up to one day of rest in-between TBI and the infusion of bone marrow may be added in this window based on logistical considerations or clinically as indicated

Bone marrow transplantation

Bone Marrow will be harvested and infused on day 0. Institutional guidelines for the infusion of bone marrow (i.e. major or minor ABO incompatible bone marrow, etc.) will be followed. The marrow infusion will be done by designated members of the BMT team. The bone marrow graft will not be manipulated to deplete T cells. The donor will be harvested with a target yield of 4 x 108 nucleated cells/kg recipient IBW. The lowest acceptable yield is 1.5 x 108 nucleated cells/kg. The CD 34+, CD4+, CD8+, and CD3+ cell count in the marrow will be quantified by flow cytometry.

Post-transplantation Cyclophosphamide

Cyclophosphamide 50mg/kg will be given on D+3 post-transplant (within 60-72 hr of marrow infusion) and on D+4 post-transplant. Cyclophosphamide will be given as an IV infusion over 1- 2 hours (depending on volume). Dosing of cyclophosphamide is based on ideal body weight for subjects whose ideal body weights less than or equal to their actual body weight. On occasion, a subject's actual body weight may be less than his/her ideal body weight, in which case cyclophosphamide will be dosed using the subject's actual body weight.

Patients will be instructed to increase fluids overnight before cyclophosphamide administration. Hydration with normal saline at 3 cc/kg/hr iv will be started 8 hr prior to cyclophosphamide, then the rate will be reduced to 2 cc/kg/hr for 1 hr pre-cyclophosphamide and continued for at least 8 hr post-cyclophosphamide or administered per institutional standards. Mesna will be given in divided doses IV 30 min pre- and at 3, 6, and 8 hours post-cyclophosphamide or administered per institutional standards. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of mesna is equal to 80% of the total daily dose of cyclophosphamide.

Patients will be instructed to increase fluids overnight before cyclophosphamide administration. Hydration will be administered per institutional standards. Protocol recommendation of normal saline at 3 cc/kg/hr iv will be started 8 hr prior to cyclophosphamide, then the rate will be reduced to 2 cc/kg/hr for 1 hr pre-cyclophosphamide and continued for at least 8 hr post-cyclophosphamide. Mesna will be administered per institutional standards. Mesna dose will be based on the cyclophosphamide dose being given. The total daily dose of mesna is equal to 80% of the total daily dose of cyclophosphamide.

It is crucial that no immunosuppressive agents are given until 24 hours after the completion of the post-transplant Cy. This includes steroids as anti-emetics.

GVHD prophylaxis

Tacrolimus On day +5, patients will begin prophylaxis with Tacrolimus (PO or IV as per institutional standards for starting this prophylaxis).Tacrolimus begins on Day 5, at least 24 hours after completion of posttransplantation Cy. The tacrolimus starting dose will be given per institutional standards for adult or pediatric patients. The recommended, but not required, The starting dose of tacrolimus is 0.015mg/kg IBW/dose IV over 4 hours every 12 hours. , or per institutional standard. Serum trough levels of tacrolimus should be measured around D+7 and the dose should be adjusted based on this level to maintain a level of 5-15 ng/ml. Tacrolimus should be converted to oral dosing when patient has a stable, therapeutic level and is able to tolerate food or other oral medications. For pediatric patients, the oral dosing is approximately two to four times the IV dosing. It is recommended that serum trough levels should be checked at steady state after any dose modification and when switching from IV to oral to ensure therapeutic trough concentrations. Serum trough concentrations should be checked at a minimum weekly thereafter and the dose adjusted accordingly to maintain a level of 5-15 ng/ml. Tacrolimus will be discontinued after the last dose on Day 90, or may be continued if active GVHD is present. This should be discussed with the PI. Tacrolimus may also be discontinued early if patients have progressive disease or relapse. If tacrolimus is stopped earlier or later than day 90 +/- 7 days , this should be discussed with the PI This should also be discussed with the PI.

Mycophenolic acid mofetil (MMF) MMF will be given at a dose of 15 mg/kg PO TID (based upon actual body weight) with the maximum total daily dose not to exceed 3 grams (1 g PO TID). MMF prophylaxis will be discontinued after the last dose on D35.

Infection prophylaxis and therapy All infection prophylaxis and therapy will be administered and discontinued as per institutional requirements. The following are recommendations only.

i) During pre-transplant evaluation patients will be screened for respiratory syncytial virus, influenza A, B and parainfluenza viruses if symptomatic. Assays of these viruses must be negative for symptomatic patients to be admitted for transplant. Strong consideration should be given to institution of ribavirin therapy if positive for adenovirus or nalidixic acid if positive for BK virus.

ii) Oral hygiene will be maintained according to institutional standards.

iii) Prophylactic anti-microbial therapy will be started during the preparative regimen, per institutional guidelines.

iv) Empiric therapy with broad-spectrum antibiotics will be instituted for the first neutropenic fever (specific agents as per current practice).

Growth factor support

Patients will receive G-CSF (Filgrastim®) 5µg/kg/d SC or IV starting at Day 5 and continuing until the ANC>1000/mm3 x 3days or two consecutive measurements over a three day period. For use in the case of fungal infections or subsequent neutropenia (ANC<500/mm3), G-CSF should be continued until the WBC>10,000-15,000.

Transfusion support Platelet and packed red cell transfusions will be given per current institutional recommendations.

Anti-ovulatory treatment Menstruating females will are recommended to should be be started on an anti-ovulatory agent, such as Lupron prior to the initiation of the preparative regimen. The treatment administered will be at the discretion of the treating physician.

Post-BMT evaluation Patients will be followed during (i) the initial post-BMT period (ii) after discharge to the referring physician as per standard practice.

ELIGIBILITY:
Presence of a suitable related HLA-haploidentical bone marrow donor.a. The donor and recipient must be identical at at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. A minimum match of 5/10 is therefore required, and will be considered sufficient evidence that the donor and recipient share one HLA haplotype.

1 year-50 years

Patients must have a confirmed histopathologic diagnosis and be classified as high risk defined by having an expected survival of < 10%. Examples include:

* Neuroblastoma or ganglioneuroblastoma

  * Failure to achieve at least a PR after induction therapy with COG ANBL0532 or standard chemotherapy
  * Refractory to induction chemotherapy with COG ANBL0532 or standard chemotherapy
  * Patients with high risk disease as defined in Appendix 1 whose autologous peripheral blood stem cell product is contaminated with neuroblastoma or who do not have an autologous product available
  * Patients with high risk disease as defined in Appendix 1 who do not meet eligibility requirements/organ function requirements for myeloablative conditioning. Patients with >5 identified lesions on the end of induction (COG ANBL0532 or standard chemotherapy) MIBG scan
* Stage 4 rhabdomyosarcoma
* Metastatic Ewing Sarcoma
* Osteosarcoma with metastatic disease beyond the lungs and/or with lung metastases not amenable to resection
* Desmoplastic small round cell tumor
* Any other solid tumor and soft tissue sarcoma with an estimated <10% chance of survival will be considered on a case by case basis at the departmental tumor board and/or sarcoma meeting

Previous therapy:

* It is expected that patients will have received upfront standard of care therapy for their respected disease
* Patients who relapse after either single or tandem autologous BMT are eligible (> 6 months must have elapsed from start of last BMT).
* Patients must be recovered from the acute toxicities of any prior chemo/radio/immunotherapy or BMT

Patients do not need to have measurable disease at time of enrollment. Patients with measurable disease must have stable disease by RECIST criteria on two scans at least 6 weeks apart.

Patients with adequate organ function as measured by

* Cardiac: Left ventricular ejection fraction at rest must be ≥ 35%, or shortening fraction > 25%.
* Hepatic: Bilirubin ≤ 3.0 mg/dL; and ALT, AST, and Alkaline Phosphatase < 5 x ULN.
* Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) > 40 mL/min/1.73m2.
* Pulmonary: FEV1, FVC, DLCO (diffusion capacity) > 50% predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation > 92% on room air.

Good performance status (Karnofsky/Lansky 60-100)

Patients (Parents/guardians for those <18) and donors must be able to sign consent forms.

Patients must be willing to participate in all stages of treatment

Criteria for recipient ineligibility Patients will not be excluded on the basis of sex, racial or ethnic background.

HIV-positive

Donor (donor anti-recipient) ABO incompatibility if an ABO compatible donor is available.

Positive leukocytotoxic crossmatch

Women of childbearing potential who currently are pregnant (HCG+) or who are not practicing adequate contraception

Uncontrolled viral, bacterial, or fungal infections.

Criteria for donor eligibility Age >0.5 years

Donors must meet the selection criteria as defined by the Foundation for the Accreditation of Hematopoietic Cell Therapy (FACT).

Lack of recipient anti-donor HLA antibody Note: In some instances, low level, non-cytotoxic HLA specific antibodies may be permissible if they are found to be at a level well below that detectable by flow cytometry. This will be decided on a case-by-case basis by the PI and one of the immunogenetics directors.

In the event that two or more eligible donors are identified, the following order of priority will be used to determine the preferred donor:

1. Medically and psychologically fit and willing to donate
2. Killer Immunoglobulin Receptor (KIR) Haplotype B Donor
3. Red blood-cell compatibility (in order of preference)

   1. RBC cross-match compatible
   2. Minor ABO incompatibility
   3. Major ABO incompatibility
4. For CMV seronegative recipients, a CMV seronegative donor. For CMV seropositive recipients, a CMV seropositive donor is preferred.
5. When possible, HLA-mismatched donors will be prioritized over HLA-matched to maximize an allogeneic benefit.

If more than one preferred donor is identified from the above list and there is no medical reason to prefer one of them, then the following guidelines are recommended:

1. If the patient is male, choose a male donor
2. Choose the youngest preferred donor
3. If the patient and family express a strong preference for a particular donor, use that one.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Shortened duration of tacrolimus as assessed by number of participants with NRM and Grade III-IV acute GVHD at Day 120 | up to 120 Days
  Safety of shortened duration immunosuppression assessed by the number of participants with non-relapse mortality (NRM) and grade III-IV acute graft versus host disease (Przepiorka criteria stages the degree of organ involvement in the skin, liver and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least sever and Stage 4+ being most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, liver 4+))

SECONDARY OUTCOMES:
Overall survival at 6 months | 6 months
  Overall survival in patients receiving reduced intensity conditioning and transplantation of partially human leukocyte antigen (HLA)-mismatched bone marrow.
Overall survival at 1 year | 1 year
  Overall survival in patients receiving reduced intensity conditioning and transplantation of partially human leukocyte antigen (HLA)-mismatched bone marrow.
Relapse | up to 2 years
  Cumulative incidence by competing risks analysis of relapse in patients receiving reduced intensity conditioning and transplantation of partially human leukocyte antigen (HLA)-mismatched bone marrow.
Non-Relapse Mortality | up to 2 years
  Time from start of intervention to death without relapse in patients receiving reduced intensity conditioning and transplantation of partially human leukocyte antigen (HLA)-mismatched bone marrow.
Event-free survival at 6 months | 6 months
  Number of months from start of intervention until first adverse event as defined as relapse/disease progression or death by CTCAE v5.0 in participants receiving reduced intensity conditioning haploBMT
Event-free survival at 1 year | 1 year
  Number of months from start of intervention until first adverse event as defined as relapse/disease progression or death by CTCAE v5.0 in participants receiving reduced intensity conditioning haploBMT
progression-free survival at 6 months | 6 months
  Number of months alive without progression in patients receiving reduced intensity conditioning and transplantation of partially human leukocyte antigen (HLA)-mismatched bone marrow.
progression-free survival at 1 year | 1 year
  Number of months alive without progression (as defined by RECIST, Any new lesion or increase of a measurable lesion by >25%; previous negative marrow positive for tumor. ** MIBG scan must be negative for patient to be classified as having a complete response. New site of disease documented by MIBG scan qualifies patient as having progressive disease.) in patients receiving reduced intensity conditioning and transplantation of partially human leukocyte antigen (HLA)-mismatched bone marrow.
acute GVHD | 30-180
  To determine the cumulative incidence by competing risks analysis of acute GVHD as defined by Przepiorka criteria stages the degree of organ involvement in the skin, liver and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least sever and Stage 4+ being most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, liver 4+)
chronic GVHD | 75days -1year
  To determine the cumulative incidence by competing risks analysis of chronic GVHD as defined by the NIH Consensus criteria

OTHER OUTCOMES:
Document toxicities | 30-180 days
  To document any unexpected toxicities after RIC haploidentical BMT.
To compare the tumor microenvironment, circulating tumor cells, and expression of MHC antigens as well as tumor specific antigens pre- and post BMT | 30days-180 days
  To compare the tumor microenvironment, circulating tumor cells, and expression of MHC antigens as well as tumor specific antigens pre- and post BMT
To document the incidence of significant viral, bacterial and fungal infections | 0-180 days
  To document the incidence of significant viral, bacterial and fungal infections as defined by the NCI's Common Terminology Criteria for Adverse Events (CTCAE) as well as the fungal criteria (proven and probable)
engraftment | day 60
  % of patients achieving donor bone marrow chimerism >/= 95% at Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Heather Symons, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Albert Einstein College of Medicine, Children's Hospital at Montefiore, The Bronx, New York
  - New York Medical Center/ Maria Fareri Children's Hospital, Valhalla, New York